CLINICAL TRIAL: NCT04114578
Title: ECHO-CDH - Exploratory Observational Prospective Study in Neonatal and Pediatric Congenital Diaphragmatic Hernia
Brief Title: Exploratory Observational Prospective Study in Neonatal and Pediatric Congenital Diaphragmatic Hernia
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gabriel Altit, Neonatologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2020-4892
Record Dates: First submitted 2019-09-27; First posted 2019-10-03 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Neonatal profile: ECHO in first 24 hours of life - ideally ECHO at Day 3-5 of life ECHO at 2-3 weeks of life or before discharge (whichever comes first) Data collected at each echocardiography: blood pressure at beginning of ECHO, pre and post-ductal saturation, respiratory support, use of inotropes and dosages, use of iNO and dosage and last blood gas
  Interventions: Other: Echocardiography
- Infant profile ( 4 month and/or 9 month): Echocardiography Age and stage questionnaires CAT/CLAMS assessment
  Interventions: Other: Echocardiography
- Pediatric profile 3, 5 and/or 8years: Echocardiography Age and stage questionnaires CAT/CLAMS assessment Results from 18 months PMA Bailey will be retrieved
  Interventions: Other: Echocardiography
- Pre-adolescent/adolescent profile 11,14 and/or 17 years: Echocardiography Pediatric Quality of Life inventory survey
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — Echocardiography has become routinely used in the diagnosis, management, and follow-up of patients with any suspected or known heart diseases. It is one of the most widely used diagnostic tests in cardiology. It can provide a wealth of helpful information, including the size and shape of the heart (internal chamber size quantification), pumping capacity, and the location and extent of any tissue damage. An echocardiogram can also give physicians other estimates of heart function, such as a calculation of the cardiac output, ejection fraction, and diastolic function (how well the heart relaxes). The acquisition usually takes about 30 minutes.

SUMMARY:
CDH is associated with lung hypoplasia, pulmonary hypertension, and left ventricular hypoplasia.

Use of new STE techniques (heart ultrasound) showed that CDH newborns have decreased LV size and function, potentially explaining the non-response to iNO, and that these cardiac findings were associated with poor outcomes. Our hypothesis: CDH newborns persist to have some degree of LV hypoplasia in the pediatric and adolescent life and pulmonary pressures remain increased during growth. Patients with decreased cardiac performance by STE and/or with PH have higher concomitant neonatal or pediatric morbidities and altered neurodevelopmental profile

DETAILED DESCRIPTION:
The principal investigator hypothesize that CDH newborns have disturbed cardiac performance and increased pulmonary pressures during neonatal life and at different pediatric ages. The principal investigator also postulate that those with decreased cardiac performance by STE and/or with PH have higher concomitant neonatal or pediatric morbidities and altered neurodevelopmental profile, that CDH patients have some remaining degree of LV hypoplasia at pediatric/adolescent age and that novel echocardiography techniques will detect anomalies not uncovered by conventional imaging.

This study is a prospective study. Cohorts will be simultaneously recruited at different neonatal and pediatric ages to create various age groups of the CDH populations.

Groups will be synchronized with the current follow-up programs to ease feasibility.

Patient Population will be CDH patients admitted to the NICU at the MCH or followed in the clinic. Patients will be recruited during hospitalization or at the different age groups corresponding to their regular CDH follow-up.

Echocardiography will be targeted to acquire: RV and LV function by STE, 3D derived RV/LV volumes and performance , conventional systolic/diastolic RV and LV function parameters (such as: ejection fraction by Simpson's Biplane, tricuspid annular plane systolic excursion and tissue Doppler velocities), cardiac outputs and pulmonary pressure estimates. For patient's safety, responsible clinician will be alerted when a clinically significant anomaly is detected on the research echocardiography. Same echocardiography protocol will be applied to controls.

Associated to echocardiography data, The principal investigator will complete a chart review to extract important neonatal/pediatric demographic and clinical data. Variables extracted, among others, will include perinatal details (mode of delivery, maternal conditions, APGAR scores), sex, birth weight, clinical course and major morbidities. Bayley Scales of Infant and Toddler Development - Third Edition, a standardized evaluation for motor, cognitive and language abilities, is done on all patients with CDH at 18 months PMA at the MCH. When available for age groups beyond 18 months of age, these scores will be recorded. As well, assessment tools describing functional and developmental status will be filled with parents (or legal guardian) and/or pre-adolescents/adolescents. These tools will be the: Ages & Stages Questionnaires 3 (a parent report of developmental skills for ages of 2 to 60 months , the Clinical Adaptive Test /Clinical Linguistic Auditory Milestone Scale (CAT/CLAMS), which has a high correlation with the Bayley Scales of Infant Development and is a neurodevelopmental assessment tool of infants and toddlers) and the Pediatric Quality of Life Inventory Survey (a pre-adolescent and adolescent report on quality of life and functional status).

Patients with CDH will be compared to controls (1:1) recruited contemporaneously. Clinics targeted for control groups include the dermatology, orthopedic, trauma follow-up and neurology clinic for benign seizures episodes.

ELIGIBILITY:
Inclusion:

* CDH patients admitted to the MCH-NICU
* CDH followed at the MCH CDH clinic

Exclusion:

* Prematurity (< 36 weeks)
* Diagnosis at > 7 days of life
* Bilateral CDH
* Congenital cardiac defect (excluding a patent ductus arteriosus (PDA), atrial septal defect (ASD) or ventricular septal defect (VSD)) and/or other major anomaly/genetic syndrome.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The control groups will be recruited in the normal nursery, in the NICU (term infants with antenatal suspicion of coarctation, which is ruled-out postnatally) or in clinics with conditions non-related to lungs or heart (such as: Inguinal hernia, Dermatology, Orthopedic and Benign Chest Pain clinics), as described in our previous published studies .
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of cardiac function | Within 24 hours of life
  Our primary outcome is cardiac function assessed by STE using peak longitudinal strain)by %
Assessment of cardiac function | Between day 3 to 5 of life
  Our primary outcome is cardiac function assessed by STE using peak longitudinal strain)by %
Assessment of cardiac function | Between 2 to 3 weeks of life
  Our primary outcome is cardiac function assessed by STE using peak longitudinal strain)by %
Assessment of cardiac function | age of 4 and/or 9 months
  Our primary outcome is cardiac function assessed by STE using peak longitudinal strain)by %
Assessment of cardiac function | 3, 5 and/or 8 years
  Our primary outcome is cardiac function assessed by STE using peak longitudinal strain)by %
Assessment of cardiac function | 11, 14 and/or 17 years
  Our primary outcome is cardiac function assessed by STE using peak longitudinal strain) by %

SECONDARY OUTCOMES:
Prevalence of pulmonary hypertension | Within 24 hours of life
  CDH newborns with pulmonary hypertension have higher concomitant neonatal or pediatric morbidities and altered neurodevelopmental profile (by mm/Hg)
Prevalence of pulmonary hypertension | Between day 3 to 5 of life
  CDH newborns with pulmonary hypertension have higher concomitant neonatal or pediatric morbidities and altered neurodevelopmental profile (by mm/Hg)
Prevalence of pulmonary hypertension | Between 2 to 3 weeks of life
  CDH newborns with pulmonary hypertension have higher concomitant neonatal or pediatric morbidities and altered neurodevelopmental profile (by mm/Hg)
Prevalence of pulmonary hypertension | age of 4 and/or 9 months
  CDH newborns with pulmonary hypertension have higher concomitant neonatal or pediatric morbidities and altered neurodevelopmental profile (by mm/Hg)
Prevalence of pulmonary hypertension | 3, 5 and/or 8 years
  CDH newborns with pulmonary hypertension have higher concomitant neonatal or pediatric morbidities and altered neurodevelopmental profile (by mm/Hg)
Prevalence of pulmonary hypertension | 11, 14 and/or 17 years
  CDH newborns with pulmonary hypertension have higher concomitant neonatal or pediatric morbidities and altered neurodevelopmental profile (by mm/Hg)

CONTACTS AND LOCATIONS:
Locations (1):
- Mcgill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No